CLINICAL TRIAL: NCT05563259
Title: The Cross-sectional and Longitudinal Study of Relationship Between Non-alcoholic Fatty Liver Disease and Cognitive Impairment
Brief Title: Cognitive Assessment and Brain Function Evaluation in Patients With Non-alcoholic Fatty Liver Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Yan Bi (Other)
Responsible Party: Sponsor-Investigator, Yan Bi, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Other Study IDs: NAFLDCOG
Record Dates: First submitted 2022-09-27; First posted 2022-10-03 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Cognitive Impairment
Keywords: MRI; cognitive function
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Groups/Cohorts Interventions Control: patients with steatosis < 5%
  Interventions: Radiation: Cognitive assessment, functional magnetic resonance imaging
- non-NASH: patients with steatosis ≥ 5% and did not achieve the criteria for NASH
  Interventions: Radiation: Cognitive assessment, functional magnetic resonance imaging
- NASH: patients with NAFLD Activity Score (NAS) ≥ 5
  Interventions: Radiation: Cognitive assessment, functional magnetic resonance imaging

INTERVENTIONS:
Radiation: Cognitive assessment, functional magnetic resonance imaging — Our study investigated cognitive function, MRI measures of brain structure and activation in patients undergoing liver biopsy. We aimed to evaluate the changes of cognition during the process of NAFLD and explore the association between brain alterations and cognition.
  Other Names: fMRI

SUMMARY:
The purpose of this study is to explore the relationship between Non-alcoholic fatty liver disease and cognitive impairment and evaluate the effect of metabolic surgery or lifestyle intervention on cognition.

DETAILED DESCRIPTION:
Previous research has shown that Non-alcoholic fatty liver disease (NAFLD) is associated with an increased risk of cognitive impairment. Even though there are many noninvasive tests available, a liver biopsy is still required for the accurate diagnosis of NAFLD. However, there are now few studies on cognitive function in patients with NAFLD based on pathological diagnosis. On one hand, in the cross-sectional study, biometric measurements, cognitive assessment, magnetic resonance imaging (MRI) results are analysed to explore the differences among control subjects and NAFLD patients undergoing liver biopsy. One the other hand, in the longitudinal study, changes in cognitive scales and MRI results in NAFLD patients both at baseline and 12-48 months after intervention are collected to investigate whether surgical intervention and weight control benefit brain function.

ELIGIBILITY:
Inclusion Criteria:

* >6 years of education
* right handed

Exclusion Criteria:

* consumed excessive alcohol (≥140 g/week for males or ≥ 70 g/week for females)
* with history of other liver diseases including chronic hepatitis, biliary obstructive diseases or autoimmune hepatitis
* with thyroid diseases
* in a state of anxiety or depression
* inability to complete cognitive function scales

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We enrolled subjects who were planning to undergo bariatric surgery in Drum Tower Hospital affiliated to Nanjing University Medical School and conducted cognitive assessment and MRI scanning within one year of biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Participants' personal information | 1 day
  Self-reported information (age in years, gender, education in years)
Physical assessments. | 1 day
  BMI (body mass index) in kg/m^2
Cognitive Assessment (MMSE) | 1 day
  Mini-Mental State Examination (MMSE) scores from 0-30, and the test means better cognition with a higher score.
Cognitive Assessment (MoCA) | 1 day
  he Montreal Cognitive Assessment (MoCA) scores from 0-30, and the test means better cognition with a higher score.
Cognitive Assessment (RBANS) | 1 day
  The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) scores from 0-800, and the test means better cognition with a higher score.
brain activation in fMRI | 1 day
  All patients underwent odor-induced task fMRI on a 3.0T MR scanner with 222 volumes for task fMRI and 230 volumes for resting-state and functional fMRI.
  The odor-induced task consisted of "fresh air" "rest" and "scent". Odor-induced brain activation was assessed by a general linear model using Statistical Parametric Mapping 12 (SPM12) software. Following extraction of the three separate conditions "fresh air," "scent," and "rest" from the whole sequence, contrasts were made for each participant between "fresh air > rest" and "scent > rest." Odor-induced fMRI data were analyzed in the mask of the olfactory network, including the regions of bilateral parahippocampus, amygdala, piriform cortex, insula, orbitofrontal cortex, hippocampus, and entorhinal cortices.

SECONDARY OUTCOMES:
Change of weight from baseline | 12-48 months
  whether body weight (kg) changes during follow-up
Change of Cognitive Assessment (MMSE) from baseline | 12-48 months
  Whether Mini-Mental State Examination (MMSE, scores from 0-30) changes during follow-up, and the test means better cognition with a higher score.
Change of Cognitive Assessment (MoCA) from baseline | 12-48 months
  Whether the Montreal Cognitive Assessment (MoCA, scores from 0-30) change during follow-up, and the test means better cognition with a higher score.
Change of Cognitive Assessment (RBANS) from baseline | 12-48 months
  Whether the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS, scores from 0-800) changes during follow-up, and the test means better cognition with a higher score.
Change of brain MRI measurement from baseline | 12-48 months
  whether brain activation changes during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- at Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No